CLINICAL TRIAL: NCT02568046
Title: An Open Label, Multi-Center Phase 1b/2a Trial Investigating Different Doses of Sym004 in Combination With FOLFIRI in Patients With Metastatic Colorectal Cancer Progressing After First-Line Therapy
Brief Title: Sym004 in Combination With FOLFIRI in Metastatic Colorectal Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued development of Sym004 in combination with FOLFIRI
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-09; 2015-003047-19 (EudraCT Number)
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — futuximab; IFL protocol; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sym004 12 mg/kg + FOLFIRI (Experimental): Phase 1b, Dose-Escalation: Dose Level 1
  Interventions: Drug: Sym004; Drug: FOLFIRI
- Sym004 9 mg/kg + FOLFIRI (Experimental): Phase 1b, Dose-Escalation: Dose Level -1
  Interventions: Drug: Sym004; Drug: FOLFIRI
- Sym004 (RP2D) + FOLFIRI (Experimental): Phase 2a, Dose-Expansion: Sym004 in the RP2D in combination with FOLFIRI
  Interventions: Drug: Sym004; Drug: FOLFIRI

INTERVENTIONS:
Drug: Sym004 — Sym004 is a 1:1 mixture of 2 monoclonal antibodies (mAbs), which bind specifically to 2 non-overlapping epitopes of the epidermal growth factor receptor (EGFR).
Drug: FOLFIRI — The standard FOLFIRI regimen consists of Irinotecan (180 mg/m^2 IV, infused over 60-90 minutes) concurrently with Folinic Acid (400 mg/m^2 IV, infused over 120 minutes) followed by 5-FU (400 mg/m^2 IV bolus, then 2400 mg/m^2 infused over 46 hours).
  Other Names: Irinotecan (Camptosar); Folinic Acid (Leucovorin); Fluorouracil (5-FU)

SUMMARY:
This is a Phase 1b/2a study investigating the safety and efficacy of Sym004, an investigational medicinal product (IMP), in combination with FOLFIRI (chemotherapy) when administered every second week (Q2W).

DETAILED DESCRIPTION:
In the Phase 1b (Dose-Escalation) portion of the trial, patients will be sequentially enrolled to dose-escalation cohorts until establishment of the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of Sym004 in combination with FOLFIRI.

The Phase 2a (Dose-Expansion) portion of the trial is expected to begin after establishing the RP2D.

Note: In January 2017, the trial was terminated during Phase 1b and enrollment was prematurely discontinued. The primary objective changed to assess the safety of the treatment combination; collection of data for secondary and exploratory objectives was omitted.

ELIGIBILITY:
Main inclusion Criteria:

1. Male or female, at least 18 years of age at the time of informed consent
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
3. Histologically or cytologically confirmed, locally advanced or metastatic colorectal cancer (CRC) that is documented to be without Kirsten rat sarcoma (KRAS) or neuroblastoma rat sarcoma (NRAS) gene mutations (i.e., tumors must express the KRAS and NRAS wild type [WT], exon 2, 3 and 4).
4. Failed (defined as radiologic progression) treatment for locally advanced or metastatic disease with first-line combination therapy of oxaliplatin and a fluoropyrimidine, with or without bevacizumab, during treatment or < 3 months after the last dose of first-line therapy and within < 3 months of C1/D1. Patients who discontinued first-line therapy due to toxicity may be enrolled provided progression occurred < 6 months after the last dose of the first-line therapy regimen.

   or Failed (defined as radiologic progression) adjuvant therapy with combination therapy of oxaliplatin and a fluoropyrimidine during treatment or within < 6 months after the last dose of oxaliplatin and within < 6 months of C1/D1.
5. Eligible for FOLFIRI
6. Measurable disease according to RECIST v1.1

Main exclusion Criteria:

1. Prior therapy with anti-EGFR antibodies, anti-EGFR small molecule inhibitors or irinotecan (CPT-11)
2. Any antineoplastic agent (standard or investigational) within 4 weeks prior to C1/D1
3. Significant gastrointestinal abnormalities
4. Patients with a significant cardiovascular disease or condition
5. Abnormal hematologic, renal or hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (8):
- United States (5):
  - UCLA School of Medicine, Los Angeles, California
  - Sharp Memorial Hosptal, San Diego, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Madrid Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled in March 2016. In January 2017, the trial was terminated early and enrollment was prematurely discontinued.
Groups:
- Dose Level 1: Sym004 12 mg/kg + FOLFIRI; Dose Level -1: Sym004 9 mg/kg + FOLFIRI: Sym004 is a 1:1 mixture of 2 monoclonal antibodies (mAbs), which bind to 2 non-overlapping epitopes of the epidermal growth factor receptor (EGFR).
  The standard FOLFIRI regimen consists of Irinotecan (180 mg/m^2 IV, infused over 60-90 minutes) concurrently with Folinic Acid (400 mg/m^2 IV, infused over 120 minutes) followed by 5-FU (400 mg/m^2 IV bolus, then 2400 mg/m^2 infused over 46 hours).
Period: Overall Study
Arm/Group | Dose Level 1: Sym004 12 mg/kg + FOLFIRI | Dose Level -1: Sym004 9 mg/kg + FOLFIRI
Started | 5 | 5
Completed (Two (2) patients were ongoing at the time of data cut-off for Primary Completion.) | 0 | 2
Not Completed | 5 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Death | 2 | 0
Not completed — Progressive Disease | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other Events | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Sym004 12 mg/kg + FOLFIRI | Dose Level -1: Sym004 9 mg/kg + FOLFIRI | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (8.55) | 61.1 (9.95) | 65.2 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5
  Spain | 2 | 3 | 5
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 170.4 (8.57) | 171.3 (4.47) | 170.9 (6.46)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 76.6 (11.97) | 82.5 (16.10) | 79.6 (13.73)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.20) | 28.0 (4.52) | 27.3 (4.19)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.9 (0.17) | 2.0 (0.24) | 1.9 (0.20)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) by Nature, Severity, and Occurrence Measured From Baseline to End of Trial Participation, as Assessed by the Common Terminology Criteria for AEs (Version 4.03) (CTCAE v4.03).
Description: AEs were coded according to the Medical Dictionary for Regulatory Activities (MedDRA) classification. The incidence and type of AEs (e.g., treatment-emergent AE [TEAE]) were summarized according to MedDRA system organ classes and preferred terms. An AE was considered as treatment-emergent if it occurred after the first treatment administration.
Time Frame: 15 months
Population: All safety analyses were conducted using the Full Analysis Set (FAS) population, defined as all patients who received at least 1 dose of trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Sym004 12 mg/kg + FOLFIRI | Dose Level -1: Sym004 9 mg/kg + FOLFIRI
Number analyzed (Participants) | 5 | 5
Participants
  At least 1 TEAE | 5 | 5
  At least 1 Serious TEAE | 3 | 2
  At least 1 Serious TEAE related to Sym004 only | 0 | 0
  At least 1 TEAE leading to Sym004 dose reduction | 1 | 2
  At least 1 TEAE leading to interruption of Sym004 | 3 | 5
  At least 1 TEAE leading to Sym004 withdrawal | 2 | 2
  At least 1 TEAE leading to FOLFIRI withdrawal | 1 | 2
  At least 1 TEAE leading to trial termination | 0 | 1
  At least 1 TEAE related to Sym004 + FOLFIRI | 4 | 3
  At least 1 TEAE related to Sym004 only | 4 | 5
  At least 1 TEAE related to FOLFIRI only | 4 | 4
  At least 1 TEAE Grade ≥3 related to Sym004+FOLFIRI | 2 | 2
  At least 1 TEAE Grade ≥ 3 related to Sym004 only | 0 | 2
  At least 1 TEAE Grade ≥ 3 related to FOLFIRI only | 1 | 1
  At least 1 dermatologic toxicity | 3 | 5
  At least 1 TEAE of hypomagnesaemia | 3 | 0
  At least 1 Infusion related reaction TEAE | 3 | 3
  At least 1 TEAE resulting in death | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse event data collection period was 15 months.
Description: Adverse event data were collected beginning with the signing of informed consent and continued through 1 month (i.e., at least 28 days) after the last administration of treatment (i.e., after both Sym004 and FOLFIRI were discontinued). After the decision was made to prematurely discontinue the trial, collection of adverse event data continued through 1 month after the last administration of Sym004.
Arm/Group | Dose Level 1: Sym004 12 mg/kg + FOLFIRI | Dose Level -1: Sym004 9 mg/kg + FOLFIRI
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5 | 2/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Sym004 12 mg/kg + FOLFIRI (N=5) | Dose Level -1: Sym004 9 mg/kg + FOLFIRI (N=5)
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Sym004 12 mg/kg + FOLFIRI (N=5) | Dose Level -1: Sym004 9 mg/kg + FOLFIRI (N=5)
Neutropenia (Blood and lymphatic system disorders) | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3
Cheilitis (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 4 | 2
Asthenia (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 0
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3
Weight decreased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated as development of Sym004 in combination with FOLFIRI was discontinued. The primary objective changed to assess the safety of the treatment combination; collection of data for secondary and exploratory objectives was omitted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications shall not disclose any Sponsor confidential information and property (not including the trial results). The Sponsor reserves the right to review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT02568046/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT02568046/SAP_001.pdf